CLINICAL TRIAL: NCT06215898
Title: Master's Thesis on the Investigation of the Effects of LSVT-BlG Protocol on Balance, Gait, Fatigue and Quality of Life in Parkinson's Patients
Brief Title: Investigation of the Effects of LSVT-BlG Protocol on Balance, Gait, Fatigue and Quality of Life in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Zeynep Ulkü Pekmezci, Physiotherapist, Izmir Bakircay University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IZBU-"PEKMEZCIZEYNEPULKU"-0001
Record Dates: First submitted 2023-12-19; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; LSVT-BIG; Balance; Gait; Fatigue; Quality of Life; Telerehabilitation; Telehealth
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Intervention Model Description: Controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients with Parkinson's Disease who were in the control group did not receive any interventional application.
- Exercise Group (LSVT-Big protocol) (Experimental): Patients with Parkinson's disease who were in the exercise group have completed a four-week supervised aerobic exercise protocol via Tele-rehabilitation.
  Interventions: Other: LSVT-BIG Group via Telerehabilitation

INTERVENTIONS:
Other: LSVT-BIG Group via Telerehabilitation — An aerobic supervised exercise protocol was implemented four times a week for four weeks in LSVT-BIG Group via a Tele-rehabilitation model.
  Arms: Exercise Group (LSVT-Big protocol)

SUMMARY:
Parkinson's disease is a progressive, degenerative neurological disease manifested by motor and non-motor symptoms. Treatment for Parkinson's disease is symptom-oriented. Treatment options include medical treatment and surgical treatment, as well as physiotherapy and rehabilitation interventions. The LSVT-BIG protocol, a physiotherapy and rehabilitation intervention, aims to overcome the insufficient speed-amplitude regulation that leads to low scaling of motion amplitude at any speed in Parkinson's disease. The protocol is applied for four weeks, four days a week, and each session is one hour. Each treatment session consists of four parts: maximal daily exercises, functional component tasks, hierarchy tasks, and grand walking. Telerehabilitation is a system established for the online delivery of different rehabilitation services via telecommunication, and it has been reported that the LSVT-BIG protocol is a viable method with image-based video conferencing systems.

This study is a randomized controlled trial designed to examine the effect of the LSVT-BIG protocol on balance, gait, fatigue and quality of life. In this direction, thirty-four Parkinson's patients will be divided into two groups by randomization method after a preliminary evaluation including balance, gait, fatigue and quality of life variables. While the telerehabilitation-based LSVT-BIG protocol was applied to the experimental group for four weeks, no physiotherapy and rehabilitation interventions would be applied to the control group in addition to the medical treatment for the same period. At the end of four weeks, both groups will be evaluated again, including balance, gait, fatigue and quality of life variables. Evaluation data will be collected from patients through face-to-face evaluation methods and prepared questionnaires and scales. The obtained data will be evaluated using appropriate statistical methods using the SPSS statistical program.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive, degenerative neurological disease manifested by motor and non-motor symptoms. Motor symptoms include resting tremor, bradykinesia, postural instability, rigidity, postural deformities, and gait disturbances. Non-motor symptoms include cognition and behavioral disorders, autonomic dysfunctions, sleep and sensory disturbances. These symptoms reduce the quality of life of patients and prevent participation in activities of daily living. Treatment for Parkinson's disease is symptom-oriented. These treatment options include medical treatment and surgical treatment, as well as physiotherapy and rehabilitation interventions.

Physiotherapy and rehabilitation interventions aim to maximize functional ability, minimize secondary complications, control unwanted side effects of medical treatment and possible motor fluctuations. For this purpose, intervention methods such as aerobic and strengthening exercises, balance and gait training, motor learning and movement strategies and the LSVT-BIG protocol are used in physiotherapy and rehabilitation programs.

LSVT-BIG protocol; derived from the Lee Silverman Voice Treatment protocol developed to improve hypophonia in Parkinson's patients, it is a treatment protocol that includes large amplitude body movements to increase both the speed and amplitude of functional movements. The goal of this protocol is to overcome the insufficient speed-amplitude regulation that leads to low scaling of the amplitude of motion at any given speed. Continuous feedback on motor performance and motion perception training in the protocol is used to offset the reduced gain in motor activities as a result of impaired sensorimotor processing. The protocol is applied for four weeks, four days a week, and each session is one hour. Each treatment session consists of four parts: maximal daily exercises, functional component tasks, hierarchy tasks, and big walking. In the study of Fishel et al., the LSVT-BIG protocol was applied to patients with intermediate Parkinson's disease. According to the results of this study, the LSVT-BIG protocol has a positive effect on balance, fall and walking variables. The study by Farley et al. showed that the LSVT-BIG protocol improved gait. It has been reported that improvement is higher especially in Hoehn Yahr stage 1 Parkinson's patients. The study by Sundaran et al suggests that balance ability in patients with Parkinson's is improved by the LSVT-BIG protocol, as assessed using the Berg Balance Scale.

Telerehabilitation is a system established for the remote delivery of different rehabilitation services via telecommunication. Online access provides advantages in terms of distance, time and cost. By taking the rehabilitation service beyond the hospital process, it allows patients to be treated in a comfortable and familiar environment. Intensive exercise programs such as the LSVT-BIG protocol impose a significant time and economic burden on patients, and there are limitations on access to the clinical setting and the practical applicability of the treatment. It is thought that these limitations can be eliminated by using the telerehabilitation method in practice. It has been reported that the LSVT-BIG protocol with telerehabilitation is a viable method with image-based video conferencing systems. The study by Fırat et al. showed that the LSVT-BIG protocol applied on the basis of telerehabilitation in Parkinson's patients gave positive results on quality of life, motor and non-motor symptoms. However, this study has some limitations such as the absence of a control group, not questioning patient satisfaction, and a small number of participants.

It is important to examine the effects of the LSVT-BIG protocol, which has been encountered in rare studies in the literature, on the motor symptoms of Parkinson's disease, since it is a current treatment approach. Few of these rare studies have used the telerehabilitation method despite the advantages it provides. In this direction, this study was planned to examine the effect of LSVT-BIG protocol applied on the basis of telerehabilitation on balance, gait, fatigue and quality of life in Parkinson's patients.

Thirty-four Parkinson's patients will be included in the study. After the first evaluation, the patients included in the study will be divided into two groups, defined as the experimental and control groups, by randomization method. The telerehabilitation-based LSVT-BIG protocol will be applied to the experimental group for four weeks, four times a week and each session for one hour, accompanied by a physiotherapist and with one-on-one participation. The control group will not be included in any physiotherapy and rehabilitation practices in addition to their basic medical treatments during this period. At the end of four weeks, a final evaluation will be made for both groups. Evaluation data will be collected from patients through face-to-face evaluation methods, questionnaires and scales.

Demographic characteristics of the patients (gender, age, height, body weight, body mass index, duration of the disease, dominant side, occupation, marital status, history, family history and medications used), Hoehn Yahr Stage and UPDRS Score will be recorded. Activity-Specific Balance Confidence Scale and Berg Balance Scale will be used for balance assessment. In addition, one-leg standing test will be applied for the evaluation of static balance and the four-step square test will be applied for the evaluation of dynamic balance. For gait assessment, Dynamic Gait Index and Figure of 8 Walk Test will be applied. Parkinson's Fatigue Scale-16 will be used for fatigue assessment and Parkinson's Disease Questionnaire-8 will be used for quality of life assessment. Telehealth Satisfaction Questionnaire will be applied in order to evaluate the satisfaction of the patient with the physiotherapy and rehabilitation approach applied to the experimental group.

The data obtained will be analyzed using the "Statistical Package for Social Sciences (SPSS)" statistical program.

ELIGIBILITY:
Inclusion Criteria:

* Have had Parkinson's Disease
* Grade 1-3 on the Hoehn-Yahr Scale
* Stability of drug therapy taken in the last month
* Being in the "ten" period of the patients
* Volunteer to participate in the study

Exclusion Criteria:

* Having other neurological, cardiovascular, or orthopedic disorder that may impair mobility have serious hearing and vision problems
* Having an additional neurological or psychiatric illness
* Not having the appropriate equipment for telerehabilitation sessions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Berg Balance Assessment | 4 weeks
  Patients' balance was assessed with Berg Balance Scale
Four Step Square Test | 4 weeks
  Four Step Square Test was used to assess patients' balance.

SECONDARY OUTCOMES:
Demographic data form | 4 weeks
  Information were gathered via a simple data form.
Dynamic gait index evaluation | 4 weeks
  Patients' walking capabilities were evaluated via "Dynamic walking index "
Assesment of quality of life | 4 weeks
  Patients' quality of life was assessed with PQOL-8 questionnaire.Minimum and maximum scores are between 1 and 29,respectively.
Fatigue assessment | 4 weeks
  Patients' fatigue level was assessed with Parkinson Fatigue Questionnaire.Minimum and maximum scores are between 16 and 80,respectively.
Assessment of the severity of Parkinson's disease | 4 weeks
  Patients' fatigue level was assessed with Unified Parkinson's Disease Rating Scale (UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Alper Tuğral, Ph.D., Study Director — Izmir Bakircay University
Locations (1):
- Bakircay University, Izmir, Turkey (Türkiye)